CLINICAL TRIAL: NCT06109116
Title: Effects of Self-myofascial Release on Hamstring Flexibility in Patients With Non Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sana REC-01679
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Nonspecific Low Back Pain
Keywords: Hamstring flexibility; Non specific low back pain; Self myofascial release

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self myofascial release + Conventional PT (Experimental): The participant will be asked to sit on a chair and feet resting on the ground. A tennis ball is used on the sole of each foot behind the metatarsal heads to the heel concentrating on the medial arch for 2 minutes in sitting position, with as much pressure as they could, pushing into discomfort but not pain. Frequency: 3 times/week for 3 weeks Intensity: moderate intensity (pain free) Time: 35 mins Type: Self myofascial release to improve hamstring flexibility Conventional PT including Hot pack, Knee to chest exercise, bridging exercise, Straight leg raise exercise, Ankle pumping exercise, Superman position exercise.
  .
  Interventions: Other: Self myofascial release+ Conventional PT
- Conventional PT (Other): Hot pack, Knee to chest exercise, Bridging exercise, Straight leg raise exercise, Ankle pumping exercise, Superman position exercise Frequency: 3 times/week for 3 weeks Intensity: moderate intensity (pain free) Time: 30 mins Type: Self myofascial release to improve hamstring flexibility
  Interventions: Other: Conventional PT

INTERVENTIONS:
Other: Self myofascial release+ Conventional PT — The participant will be asked to sit on a chair and feet resting on the ground. A tennis ball is used on the sole of each foot behind the metatarsal heads to the heel Conventional PT including Hot pack,Knee to chest exercise, Bridging exercise, Straight leg raise exercise, Ankle pumping exercise, Superman position exercise concentrating on the medial arch for 2 minutes in sitting position,with as much pressure as they could, pushing into discomfort but not pain Frequency: 3 times/week for 3 weeks Intensity: moderate intensity (pain free) Time: 35 mins Type: Self myofascial release to improve hamstring flexibility
  Arms: Self myofascial release + Conventional PT
Other: Conventional PT — Hot pack,Knee to chest exercise, Bridging exercise, Straight leg raise exercise, Ankle pumping exercise, Superman position exercise .
  Frequency: 3 times/week for 3 weeks Intensity: moderate intensity (pain free) Time: 30 mins
  Arms: Conventional PT

SUMMARY:
The aim of this preliminary study suggest the addition of self myofascial release to a therapeutic exercise program in reducing hamstring flexibility and would have additional effects on decreasing pain intensity in individuals with non specific low back pain.

DETAILED DESCRIPTION:
There are different treatments that can affect the facial tissue, but MFR techniques have shown promising effects in reducing pain, improving flexibility and daily activities, these techniques involve specifically guided load long-duration mechanical forces to manipulate the myofascial complex (16). Fascia is part of a body-wide tensional force "transmission system" as facial system is innervated by mechano receptors, that when manual pressure is applied may create a range of response via myofascial pathway by transmitting tensional force and decreasing muscle tension that facilitate movement and reduce pain, However in reviewing the literature, there is still theory and hypothesis in relation to the exact mechanism underlying the efficacy of facial manual therapy Self myofascial release (SMR) works under the same principle as myofascial release technique in which individual use their own body mass to exert pressure on soft tissues by tennis ball to the plantar surface of the foot and is widely used to increase flexibility and range of movement further along the posterior muscles of a proposed anatomy train.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nonspecific low back pain for at least 3 months.
* >20 degree active knee extension loss with hip in 90 degree of flexion
* NPRS >3
* Patients willing to participate and take treatment.

Exclusion Criteria:

* Patients having severe orthopedic, neurological disease
* Patients having specific diagnose cause of low back pain (infection, tumor, lumbar spine fracture, radicular pain, cauda equina syndrome)
* Involvement in regular flexibility yoga program
* Recent(<6 months) lower limb, spinal or soft tissue injuries
* Any integumentary contraindication to MFR

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Active knee extension test | 3 weeks
  Participants were lying supine on couch with both legs extended. The leg not being measured was tied with strip at mid-thigh level and the leg which was being measured was moved to 90 angle of hip flexion now participants were asked to extend knee joint as much as possible and hold for 5 second now measurements were taken by goniometer at knee joint same procedure was repeated for other leg
Numeric pain rating scale | 3 weeks
  The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale from 0 to 10. "0" = no pain and "10" = the most intense pain imaginable while the NPRS exhibited moderate reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, DPT,DSc PT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Internatinal Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No